CLINICAL TRIAL: NCT02997696
Title: A Randomised, Double-blind, Placebo Controlled, Parallel Group, Multi-centre, Study to Evaluate the Efficacy, Safety, Tolerability and Pharmacokinetics of ONO-4474 in Patients With Pain Due to Osteoarthritis of the Knee
Brief Title: A Study to Evaluate ONO-4474 in Patients With Pain Due to Osteoarthritis of the Knee
Acronym: MOTION
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was stopped for business reasons. No safety issues were reported.
Sponsor: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ONO-4474-02; 2016-002675-97 (EudraCT Number)
Record Dates: First submitted 2016-12-02; First posted 2016-12-20 (Estimated); Last update posted 2018-02-26 (Actual); Status verified 2018-02

CONDITIONS: Osteoarthritis, Knee; Pain
MeSH Terms: conditions — Osteoarthritis, Knee; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Experimental arm 1 (Experimental): ONO-4474 low dose every day for 4 weeks
  Interventions: Drug: ONO-4474
- Experimental arm 2 (Experimental): ONO-4474 high dose every day for 4 weeks
  Interventions: Drug: ONO-4474
- Placebo arm (Placebo Comparator): Placebo matching ONO-4474 every day for 4 weeks
  Interventions: Drug: Placebo matching ONO-4474

INTERVENTIONS:
Drug: ONO-4474
  Arms: Experimental arm 1; Experimental arm 2
Drug: Placebo matching ONO-4474
  Arms: Placebo arm

SUMMARY:
The purpose of this phase 2, randomised, double-blind, placebo controlled, parallel group, multicentre study is to investigate the efficacy, safety, tolerability and pharmacokinetics of a compound ONO-4474 in patients with moderate to severe pain due to osteoarthritis of the knee following 4 weeks of oral administration of ONO-4474.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic OA of the knee for ≥3 months diagnosed prior to screening as per American College of Rheumatology clinical criteria.
* Radiographic evidence of tibiofemoral OA of index knee (Kellgren-Lawrence grade 2-3), as confirmed at screening.
* Moderate to severe index knee pain due to OA requiring use of analgesic medication.
* Willing to discontinue use of all analgesic medication (aside from rescue medication) during the study.

Exclusion Criteria:

* Presence of, or history of,

  1. any inflammatory arthritis (e.g. gout, reactive arthritis, psoriatic arthritis, seronegative spondylarthropathy, septic arthritis, previous diagnosis of pseudogout in target joint with proven crystals on joint aspiration or elevated C-Reactive Protein (CRP) at time of knee arthritis flare),
  2. RPOA, osteonecrosis, osteoporotic fracture or any other painful joint disease other than OA,
  3. Secondary causes of OA; other rheumatologic or musculoskeletal conditions (e.g., rheumatoid arthritis, fibromyalgia, septic arthritis, congenital abnormality).
* Orthopaedic surgery of a lower extremity or any major surgery within the previous 6 months prior to Visit 1 or has plans for surgical intervention during the study.
* Symptomatic hip OA.
* A history of partial or complete joint replacement surgery in the index knee at any time or anticipating knee surgery during the study period.
* Significant knee injury or any knee surgery (including arthroscopy) in the index knee within 6 months prior to screening.
* Uncontrolled diabetes.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-01-09 (Actual); Study Completion 2018-01-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline in mean daily average index knee pain while walking | Week 4

SECONDARY OUTCOMES:
Safety profile assessed by adverse events, vital signs, laboratory tests, 12-lead electrocardiograms (ECG), physical examination | From baseline to study completion, an average of 6 weeks
Safety of ONO-4474 as assessed by C-SSRS (evaluation of suicidal ideation and behavior) | From baseline to study completion, an average of 6 weeks
Safety of ONO-4474 as assessed by neurological examination | From baseline to study completion, an average of 6 weeks
Change from baseline in mean daily average index knee pain while walking | Week 1, Week 2, Week 3 and Weeks 1-4
Change from baseline in Western Ontario and McMaster Universities Arthritis Index (WOMAC) pain, stiffness and physical function scores | Week 1, Week 2, Week 4 and Weeks 1-4
Change from baseline in overall WOMAC score | Week 1, Week 2, Week 4 and Weeks 1-4
Change from baseline in mean daily average index knee pain | Week 1, Week 2, Week 3, Week 4 and Weeks 1-4
Change from baseline in Patient Global Assessment | Week 1, Week 2, Week 4 and Weeks 1-4
Improvement score in Clinical Global Impression | Week 1, Week 2, Week 4 and Weeks 1-4
Change from baseline in: EuroQoL EQ-5D-5L | Week 4
Use of rescue medication as total number of tablets taken | Week 1, Week 2, Week 3, Week 4
Time to first rescue medication use | Week 4
Pharmacokinetics of ONO-4474 in plasma: Ctrough of ONO-4474 | Week 1, Week 2 and Week 4

OTHER OUTCOMES:
Percentage of patients who meet Osteoarthritis Research Society International - Outcome Measures in Rheumatology (OMERACT-OARSI) responder criteria | Week 1, Week 2 and Week 4
Percentage of patients who report a ≥30%, ≥50% or ≥70% decrease versus baseline in mean daily average index knee pain while walking | Weeks 1, 2, 3 and 4, and Weeks 1-4
Percentage of patients who report a ≥30%, ≥50% or ≥70% decrease versus baseline in WOMAC pain score | Weeks 1, 2 and 4, and Weeks 1-4
Percentage of patients who report a ≥30%, ≥50% or ≥70% decrease versus baseline in WOMAC physical function score | Weeks 1, 2 and 4, and Weeks 1-4
Change from baseline to study completion in mean daily average index knee pain while walking | From baseline to study completion, an average of 6 weeks
Change from baseline to study completion in WOMAC pain score | From baseline to study completion, an average of 6 weeks
Change from baseline to study completion in WOMAC physical function score | From baseline to study completion, an average of 6 weeks
Change from baseline to study completion in PGA | From baseline to study completion, an average of 6 weeks
Change of daily average index knee pain while walking versus daily physical activity | From baseline to study completion, an average of 6 weeks
Change of average index knee pain versus daily physical activity | From baseline to study completion, an average of 6 weeks
Ctrough versus change from baseline to Weeks 1, 2 and 4 in WOMAC pain score | Week 1, Week 2 and Week 4
Ctrough versus change from baseline to Weeks 1, 2 and 4 in WOMAC physical function score | Week 1, Week 2 and Week 4
Ctrough versus change from baseline to Weeks 1, 2 and 4 in PGA | Week 1, Week 2 and Week 4

CONTACTS AND LOCATIONS:
Overall Officials: Philip Conaghan, MBBS PhD, Principal Investigator — Leeds Institute of Rheumatic and Musculoskeletal Medicine, Chapel Allerton Hospital, Leeds, UK
Locations (47):
- Denmark (3):
  - Investigational Site, Aalborg
  - Investigational Site, Frederiksberg
  - Investigational Site 4504, Odense
- Hungary (6):
  - Investigational Site, Balatonfüred
  - Investigational Site, Budapest
  - Investigational Site, Eger
  - Investigational Site, Kistarcsa
  - Investigational Site, Mezőkövesd
  - Investigational Site, Szolnok
- Poland (19):
  - Investigational Site 4808, Bialystok
  - Investigational Site 4818, Bialystok
  - Investigational Site 4819, Bialystok
  - Investigational Site, Elblag
  - Investigational Site, Gdynia
  - Investigational Site, Katowice
  - Investigational Site, Kielce
  - Investigational Site 4810, Krakow
  - Investigational Site 4812, Krakow
  - Investigational Site, Lublin
  - Investigational Site, Nadarzyn
  - Investigational Site, Poznan
  - Investigational Site, Siedlce
  - Investigational Site, Staszów
  - Investigational Site 4811, Warsaw
  - Investigational Site 4815, Warsaw
  - Investigational Site, Wroclaw
  - Investigational Site 4801, Zamość
  - Investigational Site 4816, Zamość
- Spain (10):
  - Investigational Site, A Coruña
  - Investigational Site 3406, Barcelona
  - Investigational Site 3407, Barcelona
  - Investigational Site 3402, Madrid
  - Investigational Site 3410, Madrid
  - Investigational Site, Móstoles
  - Investigational Site, Sabadell
  - Investigator Site, Santiago de Compostela
  - Investigational Site, Seville
  - Investigational site, Villajoyosa
- United Kingdom (9):
  - Investigational Site, Barnsley
  - Investigational Site, Blackpool
  - Investigational Site 4401, Leeds
  - Investigational Site 4410, Leeds
  - Investigational Site, Liverpool
  - Investigational Site, Manchester
  - Investigational Site, Middlesex
  - Investigational Site, North Shields
  - Investigational Site, Romford